CLINICAL TRIAL: NCT05004623
Title: Early Feasibility Study of an Open-Field Handheld Wireless Fluorecence Imaging System for Detection of Sentinel Lymph Nodes in Women With Cervical and Uterine Cancers
Brief Title: Early Feasibility Study of the "Easy Light" Fluorecence Imaging System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Responsible Party: Principal Investigator, Thales Paulo Batista, Consulting, Professor Fernando Figueira Integral Medicine Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 45814621.5.0000.5201
Record Dates: First submitted 2021-06-16; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Uterine Cervical Neoplasms; Uterine Neoplasms
Keywords: Sentinel Lymph Node Biopsy; Fluorescence; Indocyanine Green
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: This is an early feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sentinel Lymph Node Biopsy (Other): Sentinel lymph node biopsy by indocyanine green (ICG) fluorescent dye technique, using a prototype of the Easy Light device. Lymph node dissection in each hemipelvis should be performed as standard if no sentinel lymph node is detected. Decision of proceeding with complementary lymph node dissection after sentinel lymph node detection is a surgeon decision, according to his/her usual practice.
  Interventions: Device: Sentinel Lymph Node Biopsy

INTERVENTIONS:
Device: Sentinel Lymph Node Biopsy — Detection of sentinel lymph nodes by indocyanine green (ICG) fluorescent dye technique, using a prototype of the Easy Light device.

SUMMARY:
This is an early feasibility study to evaluate the device functionality of an open-field handheld wireless fluorecence imaging system for detection of sentinel lymph nodes in women with cervical and uterine cancers who underwent open surgery.

DETAILED DESCRIPTION:
This study was designed to clinically evaluate the functionality of an prototype of our near-infrared fluorescence device named Easy Light. In brief, this device is an open-field handheld wireless fluorecence imaging system that allows real-time visualization of fluorescent dyes such as indocyanine green (ICG) using smartphones and tablets. The handheld is a rechargeable device responsible for excitation of the operative field with infra-red lighting and for capturing the fluorescence emitted by de fluorescent dye to be visualized via wi-fi in the smartphones and tablets using a pre-installed application software. Following the standards of near-infrared fluorescence for detection of sentinel lymph nodes in gynecological malignancies, the hypothesis was the identification of sentinel lymph nodes after lymphatic mapping by interstitial indocyanine green injection in the cervix was feasible with the use of our device named Easy Light.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy-proven cervical or uterine cancers;
2. Clinical stage I or II, according to FIGO - The International Federation of Gynecology and Obstetrics;
3. Indication for sentinel lymph node biopsy with or without complementary lymphadenectomy by her medical assistant;
4. Performance status of 0-2;
5. No synchronous malignancies or previous oncological treatments such as radiation or major abdominal surgery;
6. Absence of neuro-psychiatric disorders, apparent or confirmed infections, history of drug allergies, limiting obesity for surgery, and pregnancy or breast feeding;
7. Appropriated cardio-respiratory, hepato-renal and hematological reserves;
8. Signing of the Consent Form.

Exclusion Criteria:

1. Perioperative impossibility to inject the fluorescent dye indocyanine green in the cervical region due to any locorregional reason.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
The ability to detect sentinel lymph nodes. | Intraoperativelly
  The ability to detect at least one sentinel lymph node per patient during open surgeries.

CONTACTS AND LOCATIONS:
Overall Officials: Thales P Batita, PhD, Principal Investigator — IMIP, Department of Surgery/Oncology
Locations (1):
- IMIP - Instituo de Medicina Integral Professor Fernando Figueira, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No